CLINICAL TRIAL: NCT02665468
Title: eHealth Partnered Evaluation Initiative (PEC 15-470)
Brief Title: eHealth Partnered Evaluation Initiative
Acronym: eHealth PEI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PEX 16-001; PEC 15-470 (Other Grant/Funding Number: QUERI Partnered Evaluation Center)
Record Dates: First submitted 2016-01-05; First posted 2016-01-27 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2018-01

CONDITIONS: Non-secure Message Senders
Keywords: Supported adoption; Secure messaging; Patient aligned care team (PACT); My HealtheVet Coordinator

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Supported Adoption Intervention (SAI) (Other): Supported adoption intervention
  Interventions: Behavioral: Supported adoption intervention
- Arm 2: General wellness information (Active Comparator): General wellness information
  Interventions: Behavioral: Active comparator control

INTERVENTIONS:
Behavioral: Supported adoption intervention — An intervention where a healthcare system implements quality improvement by sending patients proactive reminders, motivational messages, and educational support to encourage use of a new service (i.e., secure messaging)
  Other Names: SAI
  Arms: Arm 1: Supported Adoption Intervention (SAI)
Behavioral: Active comparator control — The investigators will use an attention control (a control intended to balance the attention Veterans receive from the facility mailings and to enhance masking of intervention versus control). As an attention control must not have information about the intended intervention, the investigators will mail out general wellness information available on the VHA National Center for Prevention
  Other Names: General wellness information
  Arms: Arm 2: General wellness information

SUMMARY:
On October 1, 2016, the VHA Office of Telehealth and the Connected Health Office will merge to create a single entity that will be responsible for the implementation and evaluation of eHealth technologies across the healthcare system. In an effort to successfully fulfill its mission, the new combined Connected Health/Telehealth Office is pledging $1,100,000 for an eHealth Partnered Evaluation Initiative (PEI) to support the further implementation of eHealth technologies across VHA, and to measure their impacts on dimensions of access and other outcomes. Developed in close consultation with leadership of the new office, the proposed objectives of the eHealth PEI are to (1) implement a patient-level "supported adoption intervention" for secure messaging and evaluate the impact of secure messaging use through a rapid, one-year randomized trial; and (2) evaluate the initial rollout of VHA's automated telehealth text messaging system to Veterans and clinical team members.

DETAILED DESCRIPTION:
eHealth is a model for the delivery and receipt of healthcare services with an expanding evidence base that suggests great potential to increase access and support the transition from episodic to continuous care. In this model, patients, their families, and clinical team members use eHealth technologies that support functions (e.g., communication, behavior support, transactions) that are critical to disease prevention and health management which in turn influences behaviors, processes and outcomes.

In October 2016, the existing Office of Telehealth and the Connected Health Office will merge to create a single Office to oversee the implementation and evaluation of eHealth technologies across VHA. The new combined Connected Health/Telehealth Office will manage the full spectrum of technologies included in the current Offices of Telehealth (e.g., clinical video telehealth, home telehealth, tele-ICU) and Connected Health (e.g., patient portal, secure messaging, mobile apps), as well as new technologies that span these offices (such as the new Automated Telehealth Texting System). Recognizing the importance of rigorous evaluation to its mission, the Connected Health/Telehealth Office is pledging funds for an eHealth Partnered Evaluation Initiative (PEI) to support the further implementation of eHealth technologies across VHA, and to measure their impacts on dimensions of access, as well as Veteran and clinical team experiences, healthcare processes, and Veteran health outcomes.

Developed in close consultation with Connected Health/Telehealth Office leadership, the proposed objectives of the eHealth PEI are to (1) implement a patient-level "supported adoption intervention" for secure messaging and evaluate the impact of secure messaging use through a rapid, one-year randomized trial; and (2) evaluate the initial rollout of VHA's automated telehealth text messaging system to Veterans and clinical team members. The evaluation work associated with each of these two objectives will be guided by the Practical, Robust Implementation and Sustainability Model (PRISM).

The implementation and evaluation of eHealth technologies is not just the mission of the new Connected Health/Telehealth Office, it is also the vision of VHA. In addition to addressing the needs of the investigators' operational partner, the aforementioned objectives map to key strategies and transformational actions detailed in the Blueprint for Excellence, and align with a recently developed Virtual Access Strategy Document intended to guide the efforts of the Connected Health/Telehealth Office. The proposed eHealth PEI team includes leadership and investigators from the eHealth Quality Enhancement Research Initiative (QUERI) who are recognized authorities in informatics, implementation science, and mixed methods evaluation, and have longstanding, collaborative relationships with constituents in the Connected Health/Telehealth Office.

ELIGIBILITY:
Inclusion Criteria:

* Authenticated My HealtheVet users who have not sent a secure message
* Active patients who have an appointment scheduled in the following year

Exclusion Criteria:

* Authenticated My HealtheVet users who have sent a secure message
* Inactive patients (who do not have an appointment scheduled in the following year)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1196 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2017-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Patrick Hogan, PhD MS BS, Principal Investigator — Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA
Locations (4):
- United States (4):
  - Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA, Bedford, Massachusetts
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shimada SL, Zocchi MS, Hogan TP, Kertesz SG, Rotondi AJ, Butler JM, Knight SJ, DeLaughter K, Kleinberg F, Nicklas J, Nazi KM, Houston TK. Impact of Patient-Clinical Team Secure Messaging on Communication Patterns and Patient Experience: Randomized Encouragement Design Trial. J Med Internet Res. 2020 Nov 18;22(11):e22307. doi: 10.2196/22307. PMID 33206052
- See also: Click here for more information about this study: eHealth Partnered Evaluation Initiative (PEC 15-470) — http://www.queri.research.va.gov/partnered_evaluation/ehealth.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Supported Adoption Intervention: Supported adoption intervention
  Supported adoption intervention: An intervention where a healthcare system implements quality improvement by sending patients proactive reminders, motivational messages, and educational support to encourage use of a new service (i.e., secure messaging)
- Arm 2: Usual Care: Usual care control: As a usual control, Veterans did not receive additional information outside of usual care.
Period: Overall Study
Arm/Group | Arm 1: Supported Adoption Intervention | Arm 2: Usual Care
Started | 595 | 601
Completed | 595 | 601
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Supported Adoption Intervention | Arm 2: General Wellness Information | Total
Number analyzed (Participants) | 595 | 601 | 1196
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (13.5) | 53.8 (13.4) | 54.3 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 62 | 122
  Male | 535 | 539 | 1074
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 420 | 415 | 835
  African-American | 33 | 37 | 70
  Other Race | 6 | 5 | 11
  MIssing | 136 | 144 | 280

OUTCOME MEASURES:

1. Primary Outcome: Change in Rate of Use
Description: Measure the change in rate of use of secure messaging in intervention versus control Veterans, reported as participants in each arm that sent a secure message during study period.
Time Frame: Baseline and Six months
Population: The number of participants who received the Supported Adoption Intervention as analyzed was 2 less (these materials were returned/wrong address) than initially randomized and baseline characteristics are presented for.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Supported Adoption Intervention | Arm 2: Usual Care
Number analyzed (Participants) | 593 | 601
Participants | 85 | 28
Statistical Analysis 1: Comparison: Arm 1: Supported Adoption Intervention vs Arm 2: Usual Care; Test type: Superiority; p = 0.01, Chi-squared

2. Secondary Outcome: Patient Self-reported Access to Communication
Description: To explore the impact of secure messaging use on healthcare encounters, the investigators will compare the responses of each arm at 6-month follow-up assessment for Patient Self-reported Access to communication using 2 Questions adapted from the Survey of Healthcare Experience of Patients Scale which inquires, "How easy is it for you to communicate with your doctor when you need to?" and, "How easy is it for you to get to see your nurse when you need to?" Responses to scale were 1= "Never", 2= "Sometimes", 3= "Usually", 4= "Always"; where "Always" was the best score.
Time Frame: Six month follow-up
Population: Participants who completed the 6-month follow-up survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Supported Adoption Intervention | Arm 2: Usual Care
Number analyzed (Participants) | 269 | 316
units on a scale | 3.70 (1.11) | 3.52 (1.21)

3. Secondary Outcome: Care Coordination: Patient Assessment of Chronic Illness Care
Description: To explore the impact of secure messaging use on healthcare encounters, the investigators will use the Patient Assessment of Chronic Illness Care (PACIC) designed to assess patients' perceptions of the degree to which their care experiences are consistent with the chronic care model and includes subscale scores for patient activation, goal setting/tailoring, and follow-up/coordination. Investigators compared arms at 6-month follow-up using scale 0 (not a problem) - 4 (very big problem), where 0 indicates the desired response.
Time Frame: Six month follow-up
Population: Participants who completed 6-month follow-up assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Supported Adoption Intervention | Arm 2: Usual Care
Number analyzed (Participants) | 267 | 314
units on a scale | 2.12 (2.98) | 2.06 (2.92)

4. Secondary Outcome: Physician Accessibility and Engagement
Description: To explore the impact of secure messaging use on healthcare encounters, the investigators will compare each arm at 6-month follow-up assessment with responses from Health Care Climate Questionnaire (HCCQ), a 15-item scale adapted to assess the degree to which patient healthcare provider is accessible and supportive (taking the participant's perspective, encouraging and answering questions, supporting their plans) This is a Likert scale ranging from 1 = "Strongly Disagree" to 7 = "Strongly Agree"; where in all but one question - 1 = "Strongly Agree" is the desired response. Responses were totaled, inverting the one question and mean was determined.
Time Frame: Six months
Population: Participants who completed 6-month follow-up survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Supported Adoption Intervention | Arm 2: Usual Care
Number analyzed (Participants) | 270 | 316
units on a scale | 6.24 (1.12) | 5.97 (1.33)

ADVERSE EVENTS:
Description: All-Cause Mortality was not monitored/assessed.
Arm/Group | Arm 1: Supported Adoption Intervention | Arm 2: Usual Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/595 | 0/601
Other Adverse Events (participants affected / at risk) | 0/595 | 0/601

LIMITATIONS AND CAVEATS:
Participants were recruited at only three VA facilities, which limits generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes